CLINICAL TRIAL: NCT03080844
Title: Smoking Cessation and Brain Activation: How Practice Changes the Brain
Brief Title: Neuroimaging Studies of Practice and Smoking
Acronym: COPE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID-19
Sponsor: University of Kansas Medical Center (Other)
Collaborators: American Cancer Society, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: STUDY00004095; RSG-16-023-01 (Other Grant/Funding Number: American Cancer Society)
Record Dates: First submitted 2017-02-17; First posted 2017-03-15 (Actual); Last update posted 2021-03-05 (Actual); Status verified 2021-03

CONDITIONS: Smoking Cessation
MeSH Terms: conditions — Smoking Cessation | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Investigator
Masking Description: Primary investigator was blinded to intervention assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Practice (Experimental): Participants will be asked to delay time to smoking first cigarette of the day for up to two weeks.
  Interventions: Behavioral: Delay time to first cigarette; Behavioral: Therapy
- No Practice (Active Comparator): Participants will continue with their normal smoking behavior.
  Interventions: Behavioral: Therapy

INTERVENTIONS:
Behavioral: Delay time to first cigarette — Participants asked to delay time until they smoke first cigarette of the day.
  Arms: Practice
Behavioral: Therapy — Participants receive tips on how to resist the urge to smoke and control cravings to smoke.

SUMMARY:
The purpose of this research study is to help determine whether practicing resisting the urge to smoke changes brain function or behavior among smokers.

DETAILED DESCRIPTION:
The study is comprised of two parts: a pilot to test procedures to be used in the study, followed by the study. The pilot phase of this study will enroll 30 participants. The main study will enroll 80 after the pilot phase is completed. The pilot phase includes all of the same procedures as the main study.

ELIGIBILITY:
Inclusion Criteria:

* Smoke > 10 cigarettes per day for the last 6 months
* Smokes first cigarette within 60 minutes after waking
* Vision should be normal or corrected-to-normal (to ensure that they can accurately see the images on the screen and select the appropriate response)
* Willing to complete all appointments and change smoking behaviors for 2 weeks
* No quit attempts or attempts to cut back in the last 30 days
* No plans to quit in the next 30 days
* High school graduate or General Eduction Diploma (GED)

Exclusion Criteria:

* Serious medical illness unsuitable for the magnetic resonance imaging (MRI) scanner based on best clinical judgment
* Any neurologic or psychiatric disorder except depression, anxiety (including post-traumatic stress disorder), or attention-deficit disorder/attention-deficit hyperactivity disorder
* Currently taking anti-seizure medication
* History of concussion
* Body mass index (BMI) over 50
* Left-handedness
* History of alcohol or other substance dependence or current abuse;
* Risk for hazard due to magnetic fields such as metal in the body surgically or accidentally (e.g., pacemaker, cochlear implants, aneurysm clips, intravascular stents or coils, spinal shunt, injury involving bullets, shrapnel or metal implanted in their body, etc)
* Pregnancy

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 79 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2020-03-26 (Actual); Study Completion 2020-03-26 (Actual)

PRIMARY OUTCOMES:
Increase in percent blood oxygenation level dependent (BOLD) signal change in cognitive control network in response to smoking versus nonsmoking cues | Baseline (Day 7) to End of Study (Day 22)
  Change measured via functional magnetic resonance imaging (fMRI)

SECONDARY OUTCOMES:
Decrease in percent (BOLD) signal change in reward network in response to smoking versus nonsmoking cues | Baseline (Day 7) to End of Study (Day 22)
  Change measured via functional magnetic resonance imaging (fMRI)

CONTACTS AND LOCATIONS:
Overall Officials: Laura Martin, PhD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- Hoglund Brain Imaging Center, University of Kansas Medical Center, Kansas City, Kansas, United States

REFERENCES:
- [Derived] Fox AT, Catley D, Richter KP, Ellerbeck EF, Brucks MG, Papa VB, Martin LE. Functional brain activation changes associated with practice in delaying smoking among moderate to heavy smokers: study protocol and rationale of a randomized trial (COPE). Trials. 2018 Nov 12;19(1):623. doi: 10.1186/s13063-018-2984-x. PMID 30419931